CLINICAL TRIAL: NCT04582851
Title: Prevalence of Temporomandibular Joint Disorders Among Egyptian University Postgraduate Students
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maram Ahmed Taema, Assistant Lecturer, Cairo University
Other Study IDs: 9102020
Record Dates: First submitted 2020-10-04; First posted 2020-10-12 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postgraduate students: prevalence of TMD among postgraduate students.
  Interventions: Other: some risk factors correlated with TMD

INTERVENTIONS:
Other: some risk factors correlated with TMD — exposure factors causing TMD

SUMMARY:
The study will take place in Egypt. Postgraduate students from different faculties of the Egyptian Universities will participate. The study will begin in Decemberr 2020.

DETAILED DESCRIPTION:
Matching criteria and allocation ratio The planned study a single arm cross sectional study, in which the prevalence of students of TMD will be reported. The association between TMD and other variables will be also studied. Gender, Age, Psychological stress, non-nutritional oral habits as nail biting, lip biting, object biting and grinding of teeth (bruxism & clenching), Para-functional habits, such as intensive gum chewing, leaning of the chin on the hand and mouth breathing , previous dental treatment and previous jaw trauma will be all studied.

Data sources and management Data sources, the answered questionnaires and subsequent spread sheets will only be shared by the team members.

ddressing potential sources of bias Selection bias: Sampling will be convenient sampling, Questionnaires will be handed to the students, otherwise an email will be sent to all the students through their university email addresses if COVID-19 situation prevails.

Statistical methods Statistical methods

All confounders, effect modifiers and exposures will be controlled for by crude and adjusted regression analyses, where the primary analysis will be the adjusted one. Failure to do so as a result of violating principles of a regression model will call for a subgroup analysis, where a student t test will be used for the comparison between the subgroups.

It is also planned to study the interactions between the variables via ANOVA test if the data show normal distribution.

Participants with missing data will be excluded.

- Cross-sectional study-Since the planned sampling method is cluster sampling, where the design effect factor becomes greater than 1.

Sensitivity of the results to adjusted and crude analysis will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Postgraduate students in Egyptian universities
2. Age ranges from 18-45 years
3. Males and females

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Postgraduate students in Egyptian universities
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
prevalence of TMDs in Egyptian university students | 3 months
  by fonseca questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Diab, BDS, Principal Investigator — Cairo University; Essam Aziz, Phd, Study Chair — Cairo University; Iman Radi, PhD, Study Director — Cairo University; Maram Taema, Masters, Study Director — Cairo University; mohamed khashab, phd, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No